CLINICAL TRIAL: NCT00000941
Title: Evaluation of Potential Pharmacokinetic Interactions Between Protease Inhibitors and Lipid Lowering Agents
Brief Title: A Study on Possible Interactions Between Protease Inhibitors (Anti-HIV Drugs) and Drugs Which Lower the Level of Fat in Your Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: A5047; 10891 (Registry Identifier: DAIDS ES); ACTG A5047
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Interactions; HIV Protease Inhibitors; Ritonavir; HIV Seronegativity; Saquinavir; Nelfinavir; Anticholesteremic Agents
MeSH Terms: conditions — HIV Infections | interventions — Pravastatin; Simvastatin; Atorvastatin; Ritonavir; Nelfinavir; Saquinavir

INTERVENTIONS:
Drug: Pravastatin sodium
Drug: Simvastatin
Drug: Atorvastatin calcium
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Saquinavir

SUMMARY:
The purpose of this study is to find out whether taking protease inhibitors (anti-HIV drugs) together with lipid-lowering drugs (drugs which lower the amount of fat in the blood) has an effect on the level of drugs found in the blood compared to when these drugs are taken separately. The three protease inhibitors given in this study are ritonavir, saquinavir, and nelfinavir. The lipid-lowering drugs given are pravastatin, simvastatin, and atorvastatin.

Anti-HIV drug therapy using protease inhibitors has become very common treatment for HIV-positive patients. Recently, however, serious side effects involving how the body uses fat have been reported in people taking protease inhibitors. Examples of these side effects are redistribution of body fat and development of diabetes. People taking protease inhibitors have been found to have higher levels of fat in their blood than is normal, which can cause heart problems. It is hoped that giving lipid-lowering drugs can help prevent serious heart problems. First, however, it is important to see what happens when protease inhibitors and lipid-lowering drugs are given together.

DETAILED DESCRIPTION:
Potent antiretroviral therapy has become the standard of care for persons with HIV infection and AIDS. Recently, however, a number of complications have emerged with the widespread use of protease inhibitor (PI)-based regimens, including: hyperlipidemia, hypertriglyceridemia, diabetes mellitus, and lipodystrophy. Concern over the possibility of premature myocardial infarction has led health care providers and patients to consider treating these lipid metabolism disorders. Statin compounds have beneficial effects as lipid-lowering agents, and thereby reduce the risk of cardiovascular complications. Statin compounds such as pravastatin, simvastatin, and atorvastatin are increasingly being prescribed in persons taking PI-based potent antiretroviral therapy. It is important to determine whether there are significant drug-drug interactions between the statin compounds and PIs.

Fourteen healthy participants for each cohort of Arm A are stabilized on a fixed regimen of pravastatin (Arm A1), simvastatin (Arm A2), or atorvastatin (Arm A3) for 4 days. A baseline pharmacokinetic (PK) evaluation is completed on Day 4. Pravastatin (or simvastatin or atorvastatin) dosing stops following the Day 4 dose and PK evaluation. On Day 5, a ritonavir and saquinavir combination regimen is initiated and continued through Day 18 of the study. Pravastatin (or simvastatin or atorvastatin) dosing resumes on Day 15 and continues through Day 18. A repeat PK evaluation of pravastatin (or simvastatin or atorvastatin) in the context of combination therapy is carried out on Day 18.

Fourteen healthy participants are assigned to Arm B; these participants begin a 2-week regimen of nelfinavir. On Day 14, a baseline PK profile of nelfinavir and its M8 metabolite is carried out. Pravastatin is then added to the regimen for Days 15 to 18. On Day 18, a repeat PK evaluation of nelfinavir and the M8 metabolite is carried out in the context of combination therapy.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-negative.
* Are between the ages of 18 and 60.
* Agree to use a barrier method of birth control (e.g., a condom) during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a history of a chronic illness such as high blood pressure, heart disease, arthritis, or diabetes.
* Are pregnant or breast-feeding.
* Are taking certain medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56
Dates: Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Aweeka, Study Chair; Carl Fitchenbaum, Study Chair
Locations (13):
- United States (13):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Univ of Hawaii, Honolulu, Hawaii
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Univ of Minnesota, Minneapolis, Minnesota
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Fichtenbaum CJ, Gerber JG, Rosenkranz SL, Segal Y, Aberg JA, Blaschke T, Alston B, Fang F, Kosel B, Aweeka F; NIAID AIDS Clinical Trials Group. Pharmacokinetic interactions between protease inhibitors and statins in HIV seronegative volunteers: ACTG Study A5047. AIDS. 2002 Mar 8;16(4):569-77. doi: 10.1097/00002030-200203080-00008. PMID 11873000
- [Background] Wanke C. Pharmacokinetic interactions between protease inhibitors and statins in HIV seronegative volunteers: ACTG Study A5047, by Fichtenbaum et al. AIDS. 2003;17 Suppl 4:S109-10. No abstract available. PMID 15080191